CLINICAL TRIAL: NCT04666350
Title: Clinical Investigation Study to Evaluate the Consistency and Reproducibility of Two Consecutive Mosquito Feeding Assays in Adults With Varying Plasmodium Falciparum Gametocyte Densities
Brief Title: Clinical Investigation Study to Evaluate the Consistency and Reproducibility of Two Consecutive Mosquito Feeding Assays
Status: Completed | Type: Observational
Sponsor: PATH (Other)
Collaborators: Walter Reed Army Institute of Research (WRAIR) (U.S. Federal Agency); Kenya Medical Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: CVIA 085 -- Phase 0
Record Dates: First submitted 2020-11-24; First posted 2020-12-14 (Actual); Results first posted 2024-04-29 (Actual); Last update posted 2024-04-29 (Actual); Status verified 2022-12

CONDITIONS: Malaria
MeSH Terms: conditions — Malaria | interventions — Primaquine; Artemether, Lumefantrine Drug Combination

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Sera collected will be assayed in membrane feeding assay (risk mitigation) only if gametocyte-positive subject fails to transmit any parasites to mosquitoes in either the DSFA or DMFA performed either on day 1 or day 2. Sera will be destroyed before study close-out.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study Volunteers: Participants provided a blood sample on Day 1 for DMFA testing and then participated in the mosquito feeding assay. On Day 2 participants underwent a second DMFA and DSFA assay (within 24 hours of the first assays).
  Upon completion of Day 2 DSFA participants will receive one dose of primaquine and the first dose of a 3-day regiment of artemether/lumefantrine.
  Interventions: Other: Direct Skin Feeding Assay (DSFA); Drug: Primaquine; Drug: Artemether/Lumefantrine

INTERVENTIONS:
Other: Direct Skin Feeding Assay (DSFA) — In the direct feeding assay a cup with 60 unfed, sterile insectary-reared Anopheles gambiae mosquitoes will be allowed to feed on a participant's calf or arm for 15 minutes.
Drug: Primaquine — Participants will receive one dose of primaquine 26.3 mg tablet on Day 2 after completion of the direct feeding assay.
Drug: Artemether/Lumefantrine — Participants will receive artemether (80 mg) and lumefantrine (480 mg) combination tablets twice a day for 3 days, starting after completion of the direct feeding assay on Day 2.
  Other Names: Coartem®

SUMMARY:
The proposed trial design has been developed to assess the consistency and reproducibility of two consecutive direct skin feeding assays (DSFA) at 24-hour interval.

DETAILED DESCRIPTION:
The proposed trial design has been developed to assess the consistency and reproducibility of two consecutive direct skin feeding assays (DSFA) at 24-hour interval. The results will determine the type of pivotal trial design for a follow-on Phase 2b trial whose objective is to bridge the standard membrane feeding assay (SMFA) to the direct skin feeding assay (DSFA) and direct membrane feeding assay (DMFA) using a monoclonal antibody intervention, TB31F monoclonal antibody (mAb), which interrupts transmission from human to mosquito. The results from this experimental medicine study will inform whether the preferred "Before-After" trial design in which each human volunteer serves as their own internal control can be utilized for a follow-on Phase 2b trial.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed or thumb printed and dated informed consent form
* Stated willingness to comply with all study procedures and availability for the duration of the study
* Male or female aged between 18 years and 55 years inclusive.
* Resident within the study area
* In good general health as evidenced by medical history and clinical examination before entering the study Ability to take oral Coartem and low-dose primaquine anti-malarials upon conclusion of day 2 (2nd direct skin feed) and be willing to adhere to the medication regimen
* For females, she must be of non-childbearing potential or use appropriate measures to prevent pregnancy for 30 days after receiving Coartem and primaquine. Non-childbearing potential means she is surgically sterilized or at least one year post-menopausal. Appropriate measures to prevent pregnancy include abstinence or adequate contraceptive precautions (i.e. intrauterine contraceptive device; oral contraceptives; diaphragm or condom in combination with contraceptive jelly, cream or foam; Norplant or Depo-Provera).
* For males, he must be willing to ensure that he does not get his partner(s) pregnant for at least 3 months after treatment with primaquine. Appropriate measures to prevent pregnancy include abstinence or adequate contraceptive precautions in either the participant or the partner.
* Positive for P. falciparum gametocytes as measured by polymerase chain reaction (PCR) with cycle threshold (cT) value < 31.

Exclusion Criteria:

Presence of any signs or symptoms of malaria

* Presence of contraindications to administration of Coartem and primaquine as indicated in the respective drug package inserts
* History of severe allergic reactions to mosquito bites (other than pruritus and local swelling)
* Pregnant (i.e. a positive pregnancy test)
* Current or recent (within the preceding 2 weeks) use of antimalarial treatment
* Current participation in a malaria vaccine study
* Any other findings that the investigator feels would increase the risk of having an adverse outcome from participation in the trial.

Ages: 18 Years to 55 Years | Sex: All
Age Groups: Adult
Study Population: The target sample size for subjects with gametocytemia is approximately 45 individuals. Approximately 180 participants will be screened for gametocyte carriage by PCR to achieve the target sample size. Screening of subjects will continue until the desired sample size of gametocytemic individuals who undergo all study procedures is attained. Adults aged 18 - 55 years will be recruited from the villages in the Kombewa Health and Demographics Surveillance System (HDSS) consisting of half of Kisumu
Sampling Method: Non-Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2021-03-09 (Actual); Primary Completion 2021-12-20 (Actual); Study Completion 2021-12-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ben Andagalu, MD, Principal Investigator — Drug Resistance Laboratory, KEMRI; Hoseah Akala, MD, Principal Investigator — Drug Resistance Laboratory, KEMRI
Locations (1):
- KEMRI, Kombewa, Kenya

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Akala HM, Aponte JJ, Achola MA, Juma DW, Opot BH, Maisiba RN, Okoth RO, Juma JA, Mwakio EW, Mwalo MA, Oullo DO, Abuom D, Garges EC, Eyase FL, Tina LO, Copeland NK, Roth A, Mutunga J, Onyango I, Johnson J, Ogutu BR, Sifuna P, Hutter J, Mercer L, Raine M, Moore V, Ivinson K, Wu Y, Andagalu B, Ockenhouse CF. Consistency and reproducibility of independent feedings using blood from two consecutive days at varying Plasmodium falciparum gametocyte densities based on both direct membrane feeding assay and direct skin feeding assay. Malar J. 2025 May 16;24(1):154. doi: 10.1186/s12936-025-05360-3. PMID 40380146

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Healthy adults with no malaria symptoms were recruited from the villages in the Kombewa Health and Demographics Surveillance System (HDSS) consisting of half of Kisumu West and all of Seme Sub-Counties of Kisumu County in Kenya.
Pre-assignment Details: Four hundred participants consented and underwent screening. After informed consent was obtained participants were tested for the presence of mature stage malarial parasites (called gametocytes) in their blood. Forty-two participants met the inclusion criteria and were gametocyte positive and agreed to participate in the mosquito feeding assays.
Groups:
- Study Volunteers: Participants provided a blood sample on Day 1 for Direct Membrane Feeding Assay (DMFA) testing prior to participating in the Direct Skin Feeding Assay (DSFA). On Day 2 participants underwent the second DMFA and DSFA assay (within 24 hours of the first assays).
  Upon completion of Day 2 DSFA participants received one dose of primaquine and Coartem for 3 days.
Period: Overall Study
Arm/Group | Study Volunteers
Started | 42
Completed | 42
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Study Volunteers
Number analyzed (Participants) | 42
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.4 (9.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22
  Male | 20
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Kenya | 42
Ever had malaria? [Count of Participants; unit: Participants]
  Yes | 42
  No | 0

OUTCOME MEASURES:

1. Primary Outcome: Oocyst Prevalence
Description: Participants underwent feeding assays on two days, 24 hours apart (day 1 and Day 2). After feeding, mosquitoes were maintained in locked environmental chambers for 9 days to allow oocyst development.
  An oocyst is a structure that develops on the outer wall of the infected mosquito's stomach that contains developing sporozoites.
  Nine days after feeding mosquito midguts were dissected, stained with 1% mercurochrome and examined by optical microscopy. The number of oocysts in each midgut were recorded.
  Oocyst prevalence is defined as the percentage of mosquitoes in a cup with at least one oocyst detected in the mid-gut among the surviving mosquitoes (in the same cup) that underwent the feeding assays.
Time Frame: Feeding assays were performed on Day 1 and Day 2; Oocyst prevalence in surviving mosquitoes was assessed 9 days after feeding (Days 9 and 10).
Population: Participants with available data; one participant did not have surviving mosquitoes in any of the assays and is not included in the analysis.
  The number of mosquitoes analyzed reflects the number of surviving mosquitoes after 9 days for each feeding assay and time point.
Measure: Mean (Standard Deviation); unit: percentage of mosquitoes
Units Other Than Participants: Mosquitoes
Groups:
- Direct Skin Feeding Assay: Each participant underwent a direct skin feeding assay on Day 1 and Day 2.
- Direct Membrane Feeding Assay: Blood samples from each participant were used in a direct membrane feeding assay.
Arm/Group | Direct Skin Feeding Assay | Direct Membrane Feeding Assay
Number analyzed (Participants) | 41 | 41
Number analyzed (Mosquitoes) | 495 | 543
percentage of mosquitoes
  Day 1 Feeding Assay | 5.2 (7.8) | 6.3 (16.2)
  Day 2 Feeding Assay: number analyzed (Mosquitoes) | 467 | 476
  Day 2 Feeding Assay | 2.3 (4.9) | 2.2 (4.4)
Statistical Analysis 1: Comparison: Direct Skin Feeding Assay; Comparison of DSFA Day 2 versus Day 1. For each participant, the difference in oocyte prevalence using DSFA on Day 1 versus Day 2 was estimated. To evaluate the hypothesis that the average mean difference in the prevalence between two assays within the same subject is zero, combined estimates (weighted mean and variance) were obtained using as weight the inverse of the variance of each paired difference obtained from the Agresti and Caffo method; Test type: Other; p = 0.711, Other; The p-value is estimated assuming the combined difference over the square root of the weighted variance follows a normal distribution; Combined Difference in Prevalence = -0.025, 95% CI 2-sided [-0.160 to 0.109]
Statistical Analysis 2: Comparison: Direct Membrane Feeding Assay; Comparison of DMFA Day 2 versus Day 1. For each participant, the difference in oocyte prevalence using DMFA on Day 1 versus Day 2 was estimated. To evaluate the hypothesis that the average mean difference in the prevalence between two assays within the same subject is zero, combined estimates (weighted mean and variance) were obtained using as weight the inverse of the variance of each paired difference obtained from the Agresti and Caffo method; Test type: Other; p = 0.795, Other; [statistical method as in outcome 1, analysis 1]; Combined Difference in Prevalence = -0.016, 95% CI 2-sided [-0.139 to 0.107]

2. Secondary Outcome: Oocyst Density
Description: Participants underwent feeding assays on two days, 24 hours apart (Day 1 and Day 2). After feeding, mosquitoes were maintained in locked environmental chambers for 9 days to allow oocyst development.
  An oocyst is a structure that develops on the outer wall of the infected mosquito's stomach that contains developing sporozoites.
  Nine days after feeding mosquito midguts were dissected, stained with 1% mercurochrome and examined by optical microscopy. The number of oocysts in each midgut were recorded.
  Oocyst density is defined as the mean number of oocysts detected in infected mosquitoes that underwent feeding assays on the same participant.
Time Frame: Feeding assays were performed on Day 1 and Day 2; Oocyst density in surviving mosquitos was assessed 9 days after feeding (Days 9 and 10).
Population: Participants with available data; one participant did not have surviving mosquitoes in any of the assays and is not included in the analysis.
  The number of mosquitoes analyzed reflects the number of surviving mosquitos after 9 days for each feeding assay and time point.
Measure: Mean (Standard Deviation); unit: oocysts / mosquito
Units Other Than Participants: Mosquitoes
Arm/Group | Direct Skin Feeding Assay | Direct Membrane Feeding Assay
Number analyzed (Participants) | 41 | 41
Number analyzed (Mosquitoes) | 495 | 543
oocysts / mosquito
  Day 1 Feeding Assay | 1.1 (1.8) | 1.6 (4.1)
  Day 2 Feeding Assay: number analyzed (Mosquitoes) | 467 | 476
  Day 2 Feeding Assay | 0.4 (0.8) | 0.4 (0.8)
Statistical Analysis 1: Comparison: Direct Skin Feeding Assay; Comparison of DSFA Day 2 versus Day 1; Test type: Other; p = 0.019, Poisson Regression — Difference between days was evaluated using zero inflated Poisson regression models having as outcome the number of oocysts, as offset the number of surviving mosquitoes, and adjusted by subject; Relative Rate = 0.38, 95% CI 2-sided [0.21 to 0.70]
Statistical Analysis 2: Comparison: Direct Membrane Feeding Assay; Comparison of DMFA Day 2 versus Day 1; Test type: Other; p = 0.003, Poisson Regression — [p-value comment as in outcome 2, analysis 1]; Relative Rate = 0.23, 95% CI 2-sided [0.11 to 0.45]

3. Secondary Outcome: Sporozoite Prevalence
Description: Participants underwent feeding assays on two days, 24 hours apart (day 1 and Day 2). After feeding, mosquitoes were maintained in locked environmental chambers for 14 days to allow sporozoite development.
  Sporozoites are the forms of the plasmodium that are liberated from the oocysts in the mosquito, accumulate in the salivary glands of the mosquito, and are transferred to humans when the mosquito feeds.
  Fourteen days after feeding, salivary glands were dissected from live mosquitoes submerged in phosphate-buffered saline (PBS) in order to visualize motile sporozoites by microscopy. Sporozoite prevalence was recorded.
  Sporozoite prevalence is defined as the percentage of mosquitoes in a cup with at least one sporozoite detected in the salivary glands among the mosquitoes (in the same cup) that underwent feeding assays.
Time Frame: Feeding assays were performed on Day 1 and Day 2; Sporozoite prevalence in surviving mosquitoes was assessed 14 days after feeding (Days 14 and 15).
Population: Participants with available data; one participant did not have surviving mosquitoes in any of the assays and is not included in the analysis.
  The number of mosquitoes analyzed reflects the number of surviving mosquitos after 14 days for each feeding assay and time point.
Measure: Mean (Standard Deviation); unit: percentage of mosquitoes
Units Other Than Participants: Mosquitoes
Arm/Group | Direct Skin Feeding Assay | Direct Membrane Feeding Assay
Number analyzed (Participants) | 41 | 41
Number analyzed (Mosquitoes) | 342 | 383
percentage of mosquitoes
  Day 1 Feeding Assay | 5.1 (8.4) | 4.5 (8.0)
  Day 2 Feeding Assay: number analyzed (Mosquitoes) | 333 | 365
  Day 2 Feeding Assay | 1.8 (4.8) | 2.0 (5.7)
Statistical Analysis 1: Comparison: Direct Skin Feeding Assay; Comparison of DSFA Day 2 versus Day 1. For each participant, the difference in sporozoite prevalence using DSFA on Day 1 versus Day 2 was estimated. To evaluate the hypothesis that the average mean difference in the prevalence between two assays within the same subject is zero, combined estimates (weighted mean and variance) were obtained using as weight the inverse of the variance of each paired difference obtained from the Agresti and Caffo method; Test type: Other; p = 0.750, Other; [statistical method as in outcome 1, analysis 1]; Combined Difference in Prevalence = -0.023, 95% CI 2-sided [-0.164 to 0.118]
Statistical Analysis 2: Comparison: Direct Membrane Feeding Assay; Comparison of DMFA Day 2 versus Day 1. For each participant, the difference in sporozoite prevalence using DMFA on Day 1 versus Day 2 was estimated. To evaluate the hypothesis that the average mean difference in the prevalence between two assays within the same subject is zero, combined estimates (weighted mean and variance) were obtained using as weight the inverse of the variance of each paired difference obtained from the Agresti and Caffo method; Test type: Other; p = 0.681, Other; [statistical method as in outcome 1, analysis 1]; Combined Difference in Prevalence = -0.031, 95% CI 2-sided [-0.178 to 0.117]

4. Secondary Outcome: Sporozoite Density
Description: Sporozoite density is defined as the mean number of sporozoites detected in infected mosquitoes that underwent feeding assays.
  Due to limitation on the state of the art, it was not possible to estimate the sporozoite density using the Optical Microscopy technique.
Time Frame: Day 1 and Day 2
Population: The analysis of sporozoite density could not be conducted due to technical limitations.
Arm/Group | Direct Skin Feeding Assay | Direct Membrane Feeding Assay
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 2 days
Groups:
- Study Volunteers: Participants provided a blood sample on Day 1 for Direct Membrane Feeding Assay (DMFA) testing prior to participating in the Direct Skin Feeding Assay (DSFA). On Day 2 participants underwent the second DMFA and DSFA assay (within 24 hours of the first assays).
  Upon completion of Day 2 DSFA participants received one dose of primaquine and Coartem for 3 days, except for two women who had a positive pregnancy test at Day 2 and did not receive primaquine.
Arm/Group | Study Volunteers
All-Cause Mortality (participants affected / at risk) | 0/42
Serious Adverse Events (participants affected / at risk) | 0/42
Other Adverse Events (participants affected / at risk) | 32/42
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Study Volunteers (N=42)
Abdominal pain upper (Gastrointestinal disorders) | 1
Tonsillitis (Infections and infestations) | 1
Arthropod bite (Injury, poisoning and procedural complications) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 26
Urticaria (Skin and subcutaneous tissue disorders) | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-05-07): https://cdn.clinicaltrials.gov/large-docs/50/NCT04666350/Prot_000.pdf
  • Statistical Analysis Plan (2022-03-09): https://cdn.clinicaltrials.gov/large-docs/50/NCT04666350/SAP_001.pdf